# **Cover Page for Informed Consent Form**

| Sponsor Name | Duke Cancer Institute |
|---|---|
| NCT Number | NCT03179410 |
| Official title of Study | PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine |
| | Phenotype Prostate Cancer (PICK NEPC) |
| Document date | 03 December 2019 |

PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

#### CONCISE SUMMARY

The purpose of this study is to evaluate the safety and efficacy of a drug called avelumab in men with neuroendocrine prostate cancer. Participants will undergo a screening period that includes a physical exam, imaging scans, blood draws, and collection of archival tumor tissue. Once screening is complete, participants will come to the clinic to receive the study drug avelumab by IV infusion every 2 weeks.

During some or all of the clinic visits, participants will also be asked to complete medical exams, answer questions about any medications or adverse events, have routine imaging scans, have blood drawn for routine tests and research tests, and complete quality of life questionnaires. Participants will also be asked for permission undergo a tumor biopsy and donate some tissue to research when their cancer worsens. Participants will return to clinic 28 days after the last dose of avelumab and then be followed every 3 months for up to 3 years.

The risks for the study drug are described in this document. Some risks include: feeling tired and reactions that occur during or following the infusion which may include allergic reactions, chills, fever, muscle pain, shortness of breath, and low or high blood pressure.

If you are interested in learning more about this study, please continue to read below.

You are being asked to take part in this research study because you have neuroendocrine prostate cancer. Research studies are voluntary and include only people who choose to take part. Please read this consent form carefully and take your time making your decision. As your study doctor or study staff discusses this consent form with you, please ask him/her to explain any words or information that you do not clearly understand. We encourage you to talk with your family and friends before you decide to take part in this research study. The nature of the study, risks, inconveniences, discomforts, and other important information about the study are listed below.

Please tell the study doctor or study staff if you are taking part in another research study.

Dr. Andrew Armstrong will conduct the study and it is funded by Pfizer, Inc. Pfizer will pay Duke University to perform this research, and these funds may reimburse part of Dr. Armstrong's salary. Dr. Armstrong and one of the members of Dr. Armstrong's study team, Dr. Daniel George, have received personal compensation from Pfizer in the past for consulting or speaking engagements and may receive such compensation in the future.

#### WHO WILL BE MY DOCTOR ON THIS STUDY?

If you decide to participate, Dr. Armstrong or one of his colleagues will be your doctor for the study and will be in contact with your regular health care provider throughout the time that you are in the study and afterwards, if needed.

DUHS RB
IRB NUMBER: Pro00080869
IRB REFERENCE DATE: 12/03/2019
IRB EXPIRATION DATE: 07/06/2020

| Page 1 | of 17 |
|--------|-------|
|--------|-------|



PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

#### WHY IS THIS STUDY BEING DONE?

The purpose of this study is to evaluate the safety and efficacy of a drug called avelumab in men with neuroendocrine prostate cancer. This study will investigate how neuroendocrine prostate cancer responds to this drug and what side effects subjects experience. This study will also look different biomarkers to gain a better understanding of how avelumab affects your cancer and immune system. Biomarkers include such things as the proteins involved in tumor growth and immune system activation, circulating tumor cells (CTCs) as well as changes in your DNA. Your genes are made up of DNA. DNA is short for deoxyribonucleic acid. A gene, or DNA, contains information that determines in part the traits, such as eye color, height, or disease risk, that are passed on from parent to child. This study will determine the effect that avelumab has on these biomarkers and your tumors, both before and during the time you receive avelumab by obtaining blood samples, as well as biopsy samples.

Avelumab is an antibody (a large, Y-shaped protein used by your body's immune system to identify and neutralize foreign substances such as bacteria, viruses, and tumor cells) that affects your immune system by specifically targeting and blocking PD-L1. The PD-L1 pathway is involved in decreasing your body's natural immune response to fight cancer. By blocking PD-L1, avelumab may help your immune system stop, slow or reverse the growth of tumors. Avelumab has been approved by the Food and Drug Administration (FDA) for treatment of metastatic Merkel cell carcinoma, but it has not been approved for the treatment of neuroendocrine prostate cancer. Therefore, its use in this study is investigational. The word "investigational" means this is still being tested in research studies and is not approved by the U.S. Food and Drug Administration (FDA).

This study will take place in 2 stages. If more than 1 subject in stage 1 shows a response to the study drug, then more subjects will be enrolled in stage 2.

## HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

Approximately 23 people will take part in Stage 1 of this study at Duke and approximately 70 people will take part in both stages of this study across different hospitals and medical facilities.

#### WHAT IS INVOLVED IN THE STUDY?

If you agree to be in this study, you will be asked to sign this consent form. Before you begin the study, you will need to undergo the following tests or procedures to find out if you are eligible. Some of these tests or procedures may be part of your regular medical care and may be done even if you do not take part in the study. If you have had some of them recently, they may not need to be repeated.

- Physical exam including measurement of your weight, height and vital signs
- Complete medical history including review of prior and current medications that you are taking
- **Performance status** to evaluate how you are able to perform normal activities on a daily basis

| Subject Initials |
|------------------|
|------------------|

Form M0345



# Consent to Participate in a Research Study

PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

- Collection of blood samples (about 3 tablespoons) for routine laboratory tests (including blood cell counts, blood chemistry, and thyroid function), tests to measure your prostate-specific antigen (PSA) level and testosterone level, and tests to measure tumor markers (CEA and chromogranin A)
- **Urinalysis:** Your urine will be collected to check for signs of infection, blood, protein or sugar in your urine.
- Pathology review: You will be required to submit archival tumor tissue
- **Tumor imaging:** Your doctor will assess the status of your cancer with standard imaging techniques. These may include a bone scan and a CT/MRI of your chest, abdomen and pelvis, or a PET/CT scan.
  - O All sites of your cancer will be scanned using computed tomography (CT) or magnetic resonance imaging (MRI). A CT scan is a type of X-ray that takes images of your body with use of a small amount of radiation. An MRI is a scan that uses radio waves and a strong magnetic field to provide images of internal organs and tissues. The tumor assessment will include a scan of your chest, abdomen, and pelvis. A CT scan of your neck may also be performed if your doctor determines that it is necessary to do so. A bone scan will be done to evaluate the sites where your cancer has spread to the bone.
  - o If your study doctor determines it is necessary, you will also have a MRI scan of your brain

If eligible to participate, you will be enrolled onto the study and will begin the study visits described below.

#### **Active On-Study Phase**

During this part of the study, your study doctor will determine if you will continue receiving your standard of care treatment of androgen deprivation therapy and/or enzalutamide.

You will also begin receiving intravenous (IV) administration (using a needle placed into your vein) of the study drug avelumab every 2 weeks. One cycle lasts 4 weeks so you will receive 2 infusions per cycle.

Your doctor may prescribe you steroids or cromolyn to take prior to avelumab. These medications may reduce your risk of side effects, such as allergic reactions, while you are being give the avelumab. They may be taken by mouth (such as dexamethasone or cromolyn) or inhaled (such as cromolyn). Your doctor will tell you if taking pre-medications is appropriate for you.

In addition to the procedures listed below, you will have a bone scan and CT/MRI or a PET/CT scan every 8 weeks while you are receiving the study drug, which is the standard of care for evaluating your

| Subject Initials |
|------------------|
|------------------|



PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

type of cancer. Some of the tests or procedures listed below may also be part of your regular medical care and may be done even if you do not take part in the study.

#### Day 1 of every cycle

- Physical exam, including measurement of your weight, height and vital signs.
- Review of current medications that you are taking
- Review of any adverse events you may be experiencing
- Collection of blood samples (about 3 tablespoons) for routine laboratory tests (including blood cell counts, blood chemistry, and thyroid function), tests to measure your prostate-specific antigen (PSA) level and testosterone level, and tests to measure tumor markers (CEA and chromogranin A)
- Collection of blood samples (about 4 tablespoons) for research (cycle 1 and cycle 3 only): Several tests will be performed on the blood collected for research including but not limited to genetic sequencing and tests for biomarkers. These tests will help the researchers learn more about the effect that avelumab has on your cancer and your immune system.
- Quality of Life assessment: You will complete a questionnaire about your quality of life
  - You will complete this questionnaire on Day 1 of cycles 1, 4, 7 and every 3 subsequent cycles
- You will receive avelumab by IV infusion

## Day 15 of every cycle

- Physical exam, including measurement of your weight, height and vital signs.
- Review of current medications that you are taking
- Review of any adverse events you may be experiencing
- Collection of blood samples (about 1.5 tablespoons) for routine laboratory tests (including blood cell counts, blood chemistry)
- You will receive avelumab by IV infusion

#### **End of Study visit**

An End of Study visit will be scheduled no more than 7 days after your last dose of study drug. At this visit, the following procedures will be performed:

- Physical exam, including measurement of your weight, height and vital signs.
- Review of current medications that you are taking
- Review of any adverse events you may be experiencing

DUHS IRB
IRB NUMBER: Pro00080869
IRB REFERENCE DATE: 12/03/2019
IRB EXPIRATION DATE: 07/06/2020

PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

- Collection of blood samples (about 3 tablespoons) for routine laboratory tests (including blood cell counts, blood chemistry, and thyroid function), tests to measure your prostate-specific antigen (PSA) level and testosterone level, and tests to measure tumor markers (CEA and chromogranin A)
- Collection of blood samples (about 4 tablespoons) for research tests
  - These samples will be collected at this visit or when your cancer progresses, whichever occurs first.
- Tumor assessment using bone scan and CT/MRI scan or a PET/CT
- Quality of Life assessment

### **Optional post-progression biopsy:**

Your study doctor may determine that you will undergo a standard of care biopsy after your cancer progresses, meaning you would have the biopsy whether or not you participate in this study. The biopsy tissue may be taken from, but is not limited to, one of the following locations:

- Bone marrow
- Lymph nodes
- Liver
- Lung
- Adrenal gland

If you are having a standard of care biopsy, we would like to collect additional tissue for future research tests, including but not limited to genetic sequencing and tests for biomarkers, that will help the researchers learn more about the effect that avelumab has on your cancer and your immune system. In addition, you will be asked for permission to store tissue in the Duke Biospecimen Repository and Processing Core for future research through a separate consent form. Your study nurse will explain the details to you. If you do not want to have this biopsy or you do not want your tissue to be used for the research described in this consent form you will still be able to participate in the main clinical trial.

Please read each sentence below and think about your choice. Initial next to either "Yes" or "No" to indicate your choice. If you have any questions, please talk with your study doctor or nurse.

| | "Yes, I give my permission to collect additiona | l tissue from my | already planned | d standard of car |
|---|---|---|---|---|
| (Initial) | biopsy, if available." | | | |

"No, I do not give my permission to collect additional tissue from my already planned standard (Initial) of care biopsy."

## **Safety Follow-Up visit**

A safety follow-up visit will be scheduled about 28 days after your last dose of study drug. At this visit, the following procedures will be performed:


| DUHS | RB |
|--------|---------------------------|
| IRB NU | MBER: Pro00080869 |
| IRB RE | FERENCE DATE: 12/03/2019 |
| | PIRATION DATE: 07/06/2020 |

| Subject | Initials |
|---------|----------|



PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

- Physical exam, including measurement of your weight, height and vital signs.
- Review of current medications that you are taking
- Review of any adverse events you may be experiencing
- Collection of blood samples (about 2 tablespoons) for routine laboratory tests (including blood cell counts, blood chemistry, and thyroid function), and tests to measure your prostate-specific antigen (PSA) level and testosterone level

## **Long term Follow-up**

Following the end of your study regimen, your study doctor (or an appointed delegate) will contact you or your family or caregiver, or may access your medical records every 3 months to determine your long-term health status and to collect additional information. If you decide you no longer want to be contacted or allow access to your medical records for follow-up information, tell your study doctor.

## INFORMATION ABOUT DNA TESTING

The genetic studies described are for research purposes only. Therefore, you will receive no results from this study (except as described below). It is not the purpose of this study to look for or provide you with any medical information or diagnoses relating to your present condition or any other disease or illness. The research tests are not being used as diagnostic tests for any disease or illness. Your participation in this study is not a substitute for your regular medical care or check-ups.

Incidental findings: It is possible that this study will identify information about you that was previously unknown, such as disease status or risk. There are no plans to provide this information to you or your physician unless the information indicates that you may be at risk for a serious illness known at the time of testing to be treatable. In that case, we will attempt to notify you using the contact information you have provided, so that you can speak with Dr. Armstrong at Duke University Health System (DUHS). DUHS staff will not provide this information in a voice mail, email, or otherwise prior to contacting you. Please notify us of any change in your contact information.

| If you d | o not want to be notified of any incidental findings, please initial below. |
|---|---|
| <br>Initials | Please do not notify me of any incidental findings obtained from this research. |
| | refer, we can ask you at the time of notification whether or not you want to receive incidental information. In this case, please initial below. |
| <br>Initials | Please ask me at the time of notification whether or not I want to receive incidental findings information. |

DUHS |RB IRB NUMBER: Pro00080869 IRB REFERENCE DATE: 12/03/2019 IRB EXPIRATION DATE: 07/06/2020



PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

After providing the information to you, Dr. Armstrong may arrange for you to meet with him and/or a genetic counselor or refer you to another appropriate health care provider to review the incidental findings information with you or your physician.

<u>Use and ownership of samples:</u> By agreeing to participate in this research, you authorize DUHS, members of its staff and its business associates to use your blood and tissue for the purposes described in this consent form. DUHS will maintain these samples indefinitely or until they are exhausted.

Your blood or tissue samples may be used to generate cell lines that can be cultured and used for a longer period of time than the original samples. These cell lines will only be used as described in this consent form and will be destroyed once the research has been completed.

These samples will not be available to you for diagnostic or therapeutic purposes. Therefore, for any future diagnostic testing or treatments, a new sample will be obtained from you.

Blood and tissue collected as part of this study may be valuable for scientific, research, or teaching purposes or for the development of a new medical or commercial product. DUHS and/or the developers will assert all rights of ownership in the samples and all rights arising from use of the samples. The use of your samples may result in commercial profit. You will not be compensated for the use of your samples other than what is described in this consent form.

Availability/withdrawal of samples: You will not have access to the samples once they are obtained. Samples may be stored indefinitely. If you decide to withdraw your permission to use your samples in this research project, please contact the study doctor, Dr. Andrew Armstrong in writing and let him know you are withdrawing your permission for your identifiable samples to be stored and used for this or future research. His mailing address is DUMC Box 103861; Durham, NC 27710. At that time, we will ask you to indicate in writing if you want your unused identifiable samples destroyed or if your samples (with all identifying information removed that would link the sample to you) could be used in research. Data collected using your sample before your withdrawal will continue to be used as part of the study.

<u>Potential Risks and the Genetic Information Non-Discrimination Act (GINA):</u> There is a potential risk of loss of confidentiality. Every effort will be made to protect your confidential information, but this cannot be guaranteed. The genetic information obtained as a result of your participation in this research will not be included in your medical record. Information from which you may be personally identified will be maintained in a confidential, secure location at DUHS, accessible only by authorized members of the study team, and will not be disclosed to third parties except as described in this consent form, with your permission, or as may be required by law.

The Genetic Information Nondiscrimination Act (GINA) is a Federal law that will protect you in the following ways:

| Subject Initials |
|------------------|
|------------------|

Form M0345



# Consent to Participate in a Research Study

PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC) Investigator: Andrew Armstrong, MD, ScM

| TT 14 | 1 . | • 1 | 1 1 | 4 | , • | | | · 41 · | 1 |
|---|---|---|---|---|---|---|---|---|---|
| - Healt | n ingurance | companies and | group plans may | I not request | genetic | into | rmation t | rom this | : recearch: |
| Houn | ii iiisurance | companies and | group plans may | mot request | gonous | 11110 | i i i i a ci O i i i | TOTTI CITI | , i cocai cii, |

- Health insurance companies and group plans may not use your genetic information when making decisions regarding your eligibility or premiums;
- Employers with 15 or more employees may not use your genetic information when making a decision to hire, promote, or fire you or when setting the terms of your employment.

GINA does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA also does not protect you against discrimination based on an already-diagnosed genetic condition or disease.

Even without your name or other identifiers, your genetic information is unique to you. There is a potential risk that someone will identify you from your genetic information or learn something about you by looking at your genetic information; this risk may increase in the future as technologies advance and as more researchers study your genetic information. These risks may also affect members of your family. You should discuss your participation in this study with your family and ask the study doctor about any questions or concerns you may have.

Your samples and genetic information may be used for research for many years in the future. We will protect your privacy and confidential information by labeling your samples and genetic information only with a code number. Researchers outside of Duke University will not be given a link between the code number and your name or any other identifying information. While we hope this will prevent any potential loss of privacy or confidentiality, we cannot make any guarantees.

#### HOW LONG WILL I BE IN THIS STUDY?

You will continue to receive the study drug as long as you receive clinical benefit. This means you may also have the option to continue receiving the study drug even if your PSA level rises or your cancer appears to grow on imaging scans. Your study doctor will discuss this option with you in more detail. When you stop receiving the study drug, you will continue to be followed every 3 months (up to 3 years) for survival.

You can choose to stop participating at any time without penalty or loss of any benefits to which you are entitled. However, if you decide to stop participating in the study, we encourage you to talk to your doctor first.

## WHAT ARE THE RISKS OF THE STUDY?

Participation in a clinical trial is associated with some risks, which may include things that could make you feel unwell, uncomfortable, or harm you. You might have side effects related to the study drug while taking part in the study. Every patient taking part in the study will be closely watched for any side effects; however, the study team does not know all the effects that the study drug may have on you. These side effects may be mild or severe. In some cases, these effects might be long lasting, or permanent, and may be life threatening or in rare cases could result in death. Please refer to your study


| Subject Initials |
|------------------|
|------------------|



PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

doctor if you want to have more details on each side effect (such as expected duration, or severity). The clinical study team may give you medicines to help reduce side effects. If any of these side effects occur, you must inform your study doctor immediately.

### Risks associated with avelumab

The following side effects (considered related to study drug) have been observed in 1738 subjects who received avelumab according to the results from one oncology clinical study.

# Observed in at least 10% of subjects (10 out of 100)

- Reactions (including allergic reactions) that occur during or following infusion (may include chills, fever, muscle pain, shortness of breath, low or high blood pressure)
- Tiredness

# Observed in 2-9% of subjects (2-9 out of 100)

- Nausea
- Diarrhea
- Chills
- Reduced appetite
- Joint pain
- Fever
- Reduced function of the thyroid gland
- Itchy skin
- Vomiting
- Flu-like symptoms (including body aches, fever, and chills)
- Skin rash
- Increased blood levels of liver enzymes
- Muscle pain
- Headache
- Loss of energy

Reactions (including allergic reactions) that occur during or following the infusion (may include chills, fever, muscle pain, shortness of breath, and decrease or increase in blood pressure) are mostly mild or moderate and should resolve with a slowdown or discontinuation of the infusion and administration of medications to control the symptoms such as anti-allergic and pain-killer drugs. In some cases these reactions may be severe (less than 1% of subjects (1 out of 100)) and could require intensive medical support and even life threatening reactions may occur. During the infusion you will be observed closely for signs of an infusion reaction. The drug will be given slowly and you will also be monitored for signs of an infusion reaction for a period of time after the infusion is completed.


DUHS |RB IRB NUMBER: Pro00080869 IRB REFERENCE DATE: 12/03/2019 IRB EXPIRATION DATE: 07/06/2020



PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

You may be given drugs to reduce infusion-related reactions (side effects that occur during or following infusion) 30 to 60 minutes prior to receiving avelumab. These drugs may include, but are not limited to, antihistamines, paracetamol, steroids or cromolyn. Your study doctor or nurse will discuss which drugs you will receive and any potential side-effects.

Side effects resulting from an increased activity of the immune system have also been observed. Most of these side effects are reversible, which means they will stop once avelumab is discontinued, however in some cases these reactions may be severe (approximately 2% of subjects (2 out of 100)) and could lead to death in rare cases. The reactions that are more severe may require treatment with drugs that decrease the immune system function, also called immunosuppressant drugs (like corticosteroids or more potent drugs, such as infliximab).

The side effects resulting from an increased activity of the immune system that were observed in subjects receiving avelumab include the following:

## Observed in at least 5% of subjects (at least 5 out of 100):

- Inflammation of the thyroid gland (could include high or low function of the thyroid gland)
- Inflammation of the skin (could include skin rash, itchy skin, redness or blisters)

## Observed in 1-5% of subjects (1-5 out of 100):

- Inflammation of the large intestine (colitis)
- Inflammation of the lungs (pneumonitis)

## Observed in less than 1% of subjects (less than 1 out of 100):

- Inflammation of the liver (hepatitis)
- Decreased function of the adrenal gland (adrenal insufficiency)
- Inflammation of the muscles (myositis)
- Inflammation of the heart (myocarditis)
- Inflammation of the eyes (uveitis)

You may be given drugs to reduce infusion-related reactions (side effects that occur during or following infusion) 30 to 60 minutes prior to receiving avelumab. These drugs may include, but are not limited to, antihistamines, paracetamol (Tylenol), steroids or cromolyn.


#### Risks of antihistamines

The most common risks associated with antihistamines are:

- Dizziness
- Dry mouth, nose or throat
- Loss of coordination
- Sleepiness

| Subject | Initials |
|---------|----------|

PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

• Upset stomach (including loss of appetite, nausea, vomiting, diarrhea and constipation)

#### Risks of steroids

The most common side effects of steroids are:

- Blurred vision
- Coughing
- Changes in mood: feeling of aggression, anxiety or irritability
- Decrease in the amount of urine
- Dizziness
- Dry throat or throat irritation
- Headache
- Irregular heartbeat
- Nausea
- Numbness or tingling
- Pounding in the ears
- Rattling breathing
- Shortness of breath
- Swelling of the fingers, hands, feet or lower legs
- Trouble thinking, speaking or walking
- Weight gain

#### Risks of cromolyn

The most common side effects of cromolyn are:

- Cough
- Nasal congestion
- Nausea
- Sneezing
- Wheezing

#### Risks of paracetamol

The most common side effects of paracetamol are:

- Constipation
- Nausea
- Vomiting

#### Reproductive risks for males

Your participation in this research may damage your sperm, which could cause harm to a child that you may father while on this study. Such harm may be currently unforeseeable. If you are sexually active, you must agree to use a two medically acceptable forms of birth control (one of which must include a condom as a barrier method of contraception) in order to be in this study and for 2 months after your last

DUHS |RB IRB NUMBER: Pro00080869 IRB REFERENCE DATE: 12/03/2019 IRB EXPIRATION DATE: 07/06/2020

 Subject Initials\_\_\_\_\_



PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

dose of study drug. Medically acceptable contraceptives include: (1) surgical sterilization (such as a vasectomy), or (2) a condom used with a spermicide. Contraceptive measures such as Plan B (TM), sold for emergency use after unprotected sex, are not acceptable methods for routine use. You should inform your partner of the potential for harm to an unborn child. She should know that if pregnancy occurs, you will need to report it to the study doctor, and she should promptly notify her doctor. The study doctor will ask if your partner is willing to provide updates on the progress of the pregnancy and its outcome. If your partner agrees, this information will be provided to Pfizer, Inc. for safety monitoring follow-up.

## Risks of biopsy:

If you are already having a biopsy that is part of the regular care for your condition, obtaining additional tissue will increase the duration of your procedure. This may lead to a small increase in the chance that you will have an adverse event due to the procedure being performed.

The risks of the procedure will depend on the location of the site for biopsy. Biopsies will be performed by a radiologist under radiographic guidance. You will receive local anesthesia (numbing medication). Mild sedation in your vein may be given in some circumstances. The risks of sedation include an allergic reaction, aspiration (fluid going into the lungs), and over sedation. In addition, the IV used may cause a bruise. Rarely, an infection develops at the IV site. When the numbing medication is given, you may initially feel a burning sensation in your skin for several seconds. During the procedure, you may temporarily feel pressure and/or pain of varying degrees. If necessary, you may ask your physician for additional local anesthesia or a medication to ease your stress. You also may experience bleeding and/or bruising after the procedure is completed, and you may experience soreness in the area for a few days afterwards. Rarely, infection can develop. If you have concerns about the overall risk of your biopsy, you should discuss them with your physician.

## **Risks of Radiation:**

You will have a number of CT scans, nuclear scans and MRI scans that are part of the regular care for your condition, and you would have them whether or not you participate in this research. These studies will not add to the risk of the research. If you take part in this research and undergo a CT guided biopsy that is part of the regular care for your condition, then these studies will not add to the risk of the research. However, if you have concerns about the overall radiation exposure or MRI safety issues, you should discuss them with your physician.

## **Risks of Drawing Blood:**

Risks associated with drawing blood from your arm include momentary discomfort and/or bruising. Infection, excess bleeding, clotting, or fainting are also possible, although unlikely.

## **Drug and Food Interactions:**

For your safety, you must tell the study doctor or nurse about all the prescribed medical foods and drugs, herbal products, over-the-counter (OTC) drugs, vitamins, natural remedies, and alcohol that you are

| Sub | ject | Initials |
|-----|------|----------|



PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

taking before you start the study and before starting to take any of these products while you are on the study.

There may be risks, discomforts, drug interactions or side effects that are not yet known.

#### ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

There is no guarantee that you will receive any direct medical benefits from this study. If the study drug is effective and safe, it may help your immune system stop, slow or reverse the growth of tumors. Your overall health may improve, stay the same, or even worsen while on this study. Information from this study may help doctors learn more about avelumab and the treatment of neuroendocrine prostate cancer. This information may benefit other patients with prostate cancer or a similar condition in the future.

#### WHAT ALTERNATIVES ARE THERE TO PARTICIPATION IN THIS STUDY?

If you decide not to take part in this study, other approved treatments are available to you, which the study doctor will explain to you. You may receive treatment to control the symptoms you may be having as a result of your disease. Other options may include chemotherapy and radiation therapy. You may also choose to have no treatment for your cancer; receiving only palliative care to manage your symptoms and make you feel more comfortable. Study staff will discuss these alternative treatments and the risks and benefits associated with these treatments with you before you take part in this study.

Please talk to your doctor about these and perhaps other options.

#### WILL MY INFORMATION BE KEPT CONFIDENTIAL?

Participation in research involves some loss of privacy. We will do our best to make sure that information about you is kept confidential, but we cannot guarantee total confidentiality. Your personal information may be viewed by individuals involved in this research and may be seen by people including those collaborating, funding, and regulating the study. We will share only the minimum necessary information in order to conduct the research. Your personal information may also be given out if required by law.

In addition, your records may be reviewed in order to meet federal or state regulations. Reviewers may include representatives from the Food and Drug Administration, representatives of Pfizer, representatives of the Duke Cancer Institute, the Duke Office of Audit, Risk, and Compliance, the Duke University Health System Institutional Review Board, and others as appropriate. If any of these groups review your research record, they may also need to review your entire medical record. If this information is disclosed to outside reviewers for audit purposes, it may be further disclosed by them and may not be covered by federal privacy regulations.

Duke is participating in this study along with other member institutions of the Prostate Cancer Clinical Trial Consortium (PCCTC). As part of their reporting requirements, we will report to the PCCTC the

| Sub | ject | Initials |
|-----|------|----------|



PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

following information about all subjects that we enroll on this study: subject ID, consent date, race, and ethnicity.

As part of this study, you will be asked to have certain tests and/or procedures performed. Some of these tests and/or procedures would have been done as part of your regular care. The study doctor will use these test results both to treat you and to complete this research. These test results will be recorded in your medical record and will be reported to the research data office at Duke. Some information collected about you only for this research study may be kept in a research study record separate from your medical record, and some research information may also be part of your medical record. You will not have access to this research information until the end of the study. However, it will be available to your physicians if needed for your care.

The study results will be retained in your research record for at least six years after the study is completed. At that time either the research information not already in your medical record may be destroyed or information identifying you will be removed from such study results at DUHS. Any research information in your medical record will be kept indefinitely.

While the information and data resulting from this study may be presented at scientific meetings or published in a scientific journal, your identity will not be revealed.

Some people or groups who receive your health information might not have to follow the same privacy rules. Once your information is shared outside of DUHS, we cannot guarantee that it will remain private. If you decide to share private information with anyone not involved in the study, the federal law designed to protect your health information privacy may no longer apply to the information you have shared. Other laws may or may not protect sharing of private health information.

## WHAT ARE THE COSTS?

You or your insurance provider will be responsible and billed for all costs related to your routine medical care, including copayments and deductibles. Routine medical care services include assessments, laboratory and provider visits that you would have received for your condition if you were not participating in this research study. Not all services are covered by insurance. Some procedures or scans may require pre-authorization by your insurance plan. We will notify you if we learn that a service is not covered by your insurance plan as part of the pre-authorization process. If it is not covered, you will be responsible for paying for it. The amount of your out-of-pocket expense will depend on your insurance plan. For beneficiaries with Medicare Advantage Plans, traditional Medicare is billed for the routine cost of a research study. You may have more or higher co-pays than with a Medicare Advantage plan. Please discuss the costs of the study with your study doctor. At your request, a Financial Counselor in the clinic may provide you with an estimate of costs for routine services.

DUHS RB
IRB NUMBER: Pro00080869
IRB REFERENCE DATE: 12/03/2019
IRB EXPIRATION DATE: 07/06/2020

 Subject Initials\_\_\_\_\_



PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

The study will pay for services and procedures that are done solely for research purposes. Please talk with the PI/study team about the specific services and procedures that the study will pay for, and the ones for which you or your insurance will be responsible.

We will monitor your DUHS patient care charges to make sure that costs are directed appropriately. If you have any questions or concerns about appropriate billing, contact your study team coordinator so that he/she can help find a resolution.

Pfizer, Inc. will provide the study drug avelumab free of charge to you. Your study doctor may request that you return for a checkup before you stop your study drug if he/she thinks that stopping it suddenly may harm you and may ask you to complete the tests that would ordinarily occur when a person completes the study.

#### WHAT ABOUT COMPENSATION?

You will not receive compensation if you choose to participate in this study. However, we will provide parking vouchers to compensate for expenses related to parking.

#### WHAT ABOUT RESEARCH RELATED INJURIES?

Immediate necessary medical care is available at Duke University Medical Center in the event that you are injured as a result of your participation in this research study. However, there is no commitment by Duke University, Duke University Health System, Inc., your Duke Physicians or Pfizer, Inc. to provide monetary compensation or free medical care to you in the event of a study-related injury.

| For questions about the study or research-re | lated injury, contact Dr. Armstrong at | during |
|---|---|---|
| regular business hours and at | and ask to have Dr. Armstrong paged after hours as | nd on |
| weekends and holidays. | _ | |

# WHAT ABOUT MY RIGHTS TO DECLINE PARTICIPATION OR WITHDRAW FROM THE STUDY?

You may choose not to be in the study, or, if you agree to be in the study, you may withdraw from the study at any time. If you withdraw from the study, no new data about you will be collected for study purposes unless the data concern an adverse event (a bad effect) related to the study. If such an adverse event occurs, we may need to review your entire medical record. If your research blood sample has not already been processed for data collection, you may request that it be destroyed. Please note that it may not be possible to destroy samples, information and data created from your samples that may have already been used in research studies prior to your request.

Your samples and/or data may be stored and shared for future research without additional informed consent if identifiable private information, such as your name and medical record number, are removed. If your identifying information is removed from your samples or data, we will no longer be able to identify and destroy them.

Page 15 of

| 17 | Subject Initials |
|----|------------------|
| | - |



PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

| Your decision not to participate or to withdraw from the study will not involve any penalty or | loss of |
|---|---|
| benefits to which you are entitled, and will not affect your access to health care at Duke. If yo | ou do |
| decide to withdraw, we ask that you contact Dr. Armstrong in writing and let him know that y | ou are |
| withdrawing from the study. His mailing address is | |

We will tell you about new information that may affect your health, welfare, or willingness to stay in this study.

Your doctor may decide to take you off this study if your condition gets worse, if you have serious side effects, or if your study doctor determines that it is no longer in your best interest to continue. The sponsor or regulatory agencies may stop this study at anytime without your consent. If this occurs, you will be notified and your study doctor will discuss other options with you.

Your study doctor may ask you to return for a checkup before you stop your study drug if he or she thinks that stopping the drug suddenly may harm you.

He or she may also ask you to complete the tests that would ordinarily occur when a person completes the study.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

| For questions about the stud | y or a research-related injury, or if you | have problems, concerns, questions |
|---|---|---|
| or suggestions about the rese | earch, contact Dr. Armstrong at | during regular business |
| hours and at | and ask to have Dr. Armstrong paged | after hours and on weekends and |
| holidays. | | |

For questions about your rights as a research participant, or to discuss problems, concerns or suggestions related to the research, or to obtain information or offer input about the research, contact the Duke University Health System Institutional Review Board (IRB) Office at

DUHS RB
IRB NUMBER: Pro00080869
IRB REFERENCE DATE: 12/03/2019
IRB EXPIRATION DATE: 07/06/2020

 Subject Initials\_\_\_\_\_

Form M0345



# Consent to Participate in a Research Study

PD-L1 Inhibition as ChecKpoint Immunotherapy for NeuroEndocrine Phenotype Prostate Cancer (PICK NEPC)

Investigator: Andrew Armstrong, MD, ScM

#### STATEMENT OF CONSENT

"The purpose of this study, procedures to be followed, risks and benefits have been explained to me. I have been allowed to ask questions, and my questions have been answered to my satisfaction. I have been told whom to contact if I have questions, to discuss problems, concerns, or suggestions related to the research, or to obtain information or offer input about the research. I have read this consent form and agree to be in this study, with the understanding that I may withdraw at any time. I have been told that I will be given a signed and dated copy of this consent form."

| Signature of Subject | Date | Time |
|---------------------------------------|------|--------|
| Signature of Person Obtaining Consent | Date | - Time |